CLINICAL TRIAL: NCT04437888
Title: Randomized Blinded, Placebo Controlled Trial of Intrapoperative Ketamine for Patients Undergoing Total Joint
Brief Title: Intraoperative Ketamine for Patients Undergoing Total Joint Arthroplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Wayne E. Moschetti, Section Chief, Division of Adult Reconstructive Surgery, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D20116; STUDY02000376 (Other: Dartmouth-Hitchcock)
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Pain, Postoperative; Arthroplasty Complications
Keywords: Ketamine; Total Hip Replacement; Total Knee Replacement; Pain Catastrophizing
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, prospective double-blind, placebo controlled trial to evaluate the efficacy of intra-operative ketamine administration in patients undergoing elective total hip or knee arthroplasty, who have high pain catastrophizing scores.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigator, participant, research staff and medical provider will all be masked. The pharmacy will maintain the randomization and will provide the code at the conclusion of the study prior to data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Racemic Ketamine (Active Comparator): ketamine 0.5mg/kg bolus on induction of anesthesia and 10mcg/kg/min infusion initiated prior to incision and terminated at the completion of wound closure. Maximum ketamine dose will not exceed 500mg
  Interventions: Drug: Ketamine
- Saline (Placebo Comparator): saline in the same volume as the study drug, administered in the exact same format.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine versus saline placebo will be compared in order to evaluate the effects of Ketamine on patients that are pain catastrophizers

SUMMARY:
Prospective randomized double blinded, placebo controlled study that will evaluate the effect of intra-operative ketamine administration on post-operative analgesic requirements and self-reported pain in patients undergoing total hip and total knee arthroplasty who demonstrate high levels of pain catastrophizing.

DETAILED DESCRIPTION:
Pain management can be one of the most challenging aspects of care for total joint arthroplasty patients. Poor post-operative pain control can lead to poor patient satisfaction and functional outcomes. Moreover, prolonged post-operative opioid utilization for post-operative pain is associated with substantial adverse sequelae. Identifying patients at high risk for poor post-operative pain control, and implementing strategies to improve pain management in this population is of utmost importance. One patient feature that has been shown to reliably predict poor post-operative pain management is pain catastrophizing. Currently available self-reported metrics such as the pain catastrophizing scale allow for pre-operative identification of patients who exhibit high levels of pain catastrophizing. Furthermore, there currently exist strategies which may effectively improve post-operative pain management in this population. One such strategy is "pre-emptive" analgesia utilizing ketamine administered at the time of surgery. Ketamine is commonly utilized in the treatment of both acute and chronic pain, and is believed to reduce pain intensity through a complex mechanism involving opioid receptors and excitatory neurotransmitters. It has been utilized in a variety of surgical procedures and has consistently been shown to reduce acute post-operative pain and analgesic consumption as long as 6 months after surgery, without a significant incidence of medication related side effects. To date, no study has evaluated the use of ketamine for total joint arthroplasty patients who demonstrate high levels of pain catastrophizing. We aim to study the effect of intra-operative ketamine administration on post-operative analgesic requirements and self-reported pain in patients undergoing total hip and total knee arthroplasty who demonstrate high levels of pain catastrophizing.

ELIGIBILITY:
Inclusion Criteria:

• Adults, 18 years and older, undergoing primary total hip arthroplasty or total knee arthroplasty

Exclusion Criteria:

* History of intolerance or allergy to ketamine, either documented or self-reported.
* History of increased intra-ocular pressure, uncontrolled hypertension, increased intra-cranial pressure, psychosis.
* Unable to provide consent.
* Current incarceration.
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Total Morphine consumption during the first 48 hours post surgery | Daily for six weeks
  Morphine consumption will be measured in a pain diary for 6- weeks post-surgical procedure. Decreased is morphine consumption will indicate effectiveness of ketamine administration

SECONDARY OUTCOMES:
Hip Disability and Osteoarthritis Outcome Score for Joint Replacement (HOOS, JR.) | Pre-operation, post-operation at 6 weeks, 12 weeks, and 6 months
  six question questionnaire measuring joint specific pain and physical function, scored by summing the raw response (range 0-24) and then converting it to an interval score using the table provided below. The interval score ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health.
Knee Disability and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR.) | Pre-operation, post-operation at 6 weeks, 12 weeks, and 6 months
  Seven question questionnaire measuring joint specific pain and physical functionscored by summing the raw response (range 0-28) and then converting it to an interval score using the table provided below. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Patient-Reported Outcomes Measurement Information System (PROMIS-10) | Pre-operation, post-operation at 6 weeks, 12 weeks, and 6 months
  patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. The higher the score the healthier the subject is compared to the general population.
Pain Catastrophizing Scale (PCS) | post-operation at 6 weeks, 12 weeks, and 6 months
  The PCS is a 13 item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). The PCS is broken into three subscales being magnification, rumination, and helplessness. The higher the score, the more catastrophizing thoughts are present.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne E Moschetti, MD, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No